CLINICAL TRIAL: NCT06588829
Title: Examining the Relationship Between Burnout and Career Commitment of Occupational Therapists in Skilled Nursing Facilities
Status: Not yet recruiting | Type: Observational
Sponsor: Bay Path University (Other)
Responsible Party: Principal Investigator, Karissa Schmid, Occupational Therapist, Bay Path University
Other Study IDs: IRB # 2024_Schmid
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Burnout Among Occupational Therapists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A mixed methods cross-sectional survey was created for the proposed research questions. The survey is best for this research as it will indicate if occupational therapy practitioners (OTPs) are burnt out through the Maslach Burnout Inventory - Human Services Survey (MBI-HSS) and will provide information on a direct link to OTPs' intention of leaving or OTPs' decreased perceived quality of treatment interventions. By having clear evidence of the linkage, qualitative research generates non-numerical data to develop a deeper understanding of why OTPs are leaving the profession. By utilizing online recruitment methods, this will allow OTPs easier access and easier ability to administer. Participants will be recruited utilizing purposeful and snowball sampling techniques. Participants will be recruited from employer emails, social media and alumni pages.

Data will be collected for approximately one month, giving participants time to participate and pass along the survey to other colleagues. The survey will be completed on an anonymous online platform for ease and convenience of participation. The survey is broken into four sections. Before starting the survey, participants had to indicate that they acknowledge and accept the informed consent. If they deny the informed consent, the survey was be submitted without asking questions. Section two contained the demographic data. Section three contained the MBI-HSS. Section four included the non-standardized quantitative and qualitative questions related directly to the intention of leaving the profession and their perceived quality of treatment interventions.

Burnout is a topic that will always be around and talked about. In order to gain a better understanding of the role that burnout plays in the field of occupational therapy and the direct effects if has on therapists and the profession is important. Finding out the effects can help companies and the American Occupational Therapy Association address these issues and adjust to the current needs.

ELIGIBILITY:
Inclusion Criteria:

* Occupational Therapists or Certified Occupational Therapy Assistants Currently working in skilled nursing facilities or have worked in the last 2 years Any age range, any state Must have an active OT or COTA license

Exclusion Criteria:

* OT or COTA in a field other than skilled nursing facilities

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Occupational therapists and certified occupational therapy assistants currently working in a skilled nursing facility or have worked in a skilled nursing facility in the past two years. Participants can be any age range who hold an active license in the state they are working in.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Relationship between Burnout and Career Commitment | Baseline
Relationship between Burnout and Perceived Quality of Treatment Interventions | Baseline

IPD SHARING:
Plan to Share IPD: No